CLINICAL TRIAL: NCT02305238
Title: A Randomized, Open-label Phase 4 Study Evaluating the Efficacy and Safety of Repeated Doses of Intravitreal Aflibercept With Variable Treatment Intervals in Japanese Subjects With Neovascular Age-related Macular Degeneration
Brief Title: Japanese Treat and Extend Study of Aflibercept in Neovascular Age-related Macular Degeneration
Acronym: ALTAIR
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Bayer (Industry)
Collaborators: Regeneron Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 17668
Record Dates: First submitted 2014-11-28; First posted 2014-12-02 (Estimated); Results first posted 2018-03-12 (Actual); Last update posted 2023-11-18 (Actual); Status verified 2023-11

CONDITIONS: Wet Macular Degeneration
Keywords: Eylea,; Aflibercept; Treat and Extend regimen; Age-related macular degeneration
MeSH Terms: conditions — Wet Macular Degeneration; Macular Degeneration | interventions — aflibercept

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- 2 Weeks adjustment (Experimental): Participants received Aflibercept IVT injection at Week 0, Week 4, Week 8 and Week 16 followed by the variable treatment intervals with the criteria of Treat and Extend regimen. In the case the study eye of a participant met the criteria, the length of treatment interval was to be extended or shortened by 2 weeks from the last interval, respectively. Minimum/Maximum treatment interval is 8 weeks and 16 weeks during Week 16 to 96.
  Interventions: Drug: Aflibercept (Eylea, VEGF Trap-Eye, BAY86-5321)
- 4 Weeks adjustment (Experimental): Participants received Aflibercept IVT injection at Week 0, Week 4, Week 8 and Week 16 followed by the variable treatment intervals. In the case the study eye of a participant met the criteria of the shortening, the length of the treatment interval was to be shortened by 2 weeks. But when the last treatment interval for a participant was extended by 4 weeks from the second last interval, the treatment interval was shortened by 4 weeks. In the case the study eye of a participant met the criteria of the extension, the length of the treatment interval was to be extended by 4 weeks. But when a participant had a history of receiving treatment with interval shortened by 4 weeks during this study, the length of the extension was 2 weeks. Minimum/Maximum treatment interval is 8 weeks and 16 weeks during Week 16 to 96.
  Interventions: Drug: Aflibercept (Eylea, VEGF Trap-Eye, BAY86-5321)

INTERVENTIONS:
Drug: Aflibercept (Eylea, VEGF Trap-Eye, BAY86-5321) — Aflibercept 2mg is intravitreally injected.

SUMMARY:
To assess the efficacy of intravitreal (IVT) administration of aflibercept with two different approaches of Treat and Extend dosing regimens in Japanese subjects with neovascular (wet) Age-related Macular Degeneration (wAMD) .

To assess the safety of IVT administration of aflibercept with two different approaches of Treat and Extend dosing regimen in Japanese subjects with wAMD for up to 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Japanese men and women ≥ 50 years of age
* Active primary subfoveal choroidal neovascularization (CNV) lesions secondary to wAMD, including juxta-foveal lesions that affect the fovea as evidenced by fluorescein angiography (FA) in the study eye
* Early Treatment Diabetic Retinopathy Study (ETDRS) best-corrected visual acuity (BCVA) of 73 to 25 letters (approximately 20/40 to 20/320 at Snellen equivalent) in the study eye

Exclusion Criteria:

* Prior treatment of the study eye with intraocular anti-VEGF(Vascular Endothelial Growth Factor) agents, verteporfin photodynamic therapy (PDT), other laser, intraocular corticosteroids, surgical interventions (except cataract surgery more than 30 days prior to screening) or systemic use of anti-VEGF products within 3 months prior to study entry
* Active or suspected infection in or surrounding of the study eye
* Active severe intraocular inflammation in the study eye
* Intraocular pressure (IOP) ≥ 25 mmHg in the study eye
* Ocular condition in the study eye which may impact vision and confound study outcomes

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 288 (Actual)
Dates: Start 2014-12-19 (Actual); Primary Completion 2016-12-22 (Actual); Study Completion 2017-12-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (35):
- Japan (35):
  - Ichinomiya, Aichi-ken
  - Nagoya, Aichi-ken
  - Toyoake, Aichi-ken
  - Asahi, Chiba
  - Sakura, Chiba
  - Kōriyama, Fukushima
  - Kure, Hiroshima
  - Sapporo, Hokkaido
  - Kobe, Hyōgo
  - Inashiki-gun, Ibaraki
  - Mito, Ibaraki
  - Morioka, Iwate
  - Yokohama, Kanagawa
  - Nankoku, Kochi
  - Miyakonojō, Miyazaki
  - Iida, Nagano
  - Matsumoto, Nagano
  - Hirakata, Osaka
  - Moriguchi, Osaka
  - Sayama, Osaka
  - Takatsuki, Osaka
  - Ōtsu, Shiga
  - Chiyoda-ku, Tokyo
  - Chuoku, Tokyo
  - Hachiōji, Tokyo
  - Mitaka, Tokyo
  - Shinjuku-ku, Tokyo
  - Taito-ku, Tokyo
  - Shimonoseki, Yamaguchi
  - Ube, Yamaguchi
  - Chūō, Yamanashi
  - Fukuoka
  - Miyazaki
  - Okayama
  - Osaka

REFERENCES:
- [Result] Okada AA, Takahashi K, Ohji M, Moon SC, Machewitz T, Sasaki K; ALTAIR Study Investigators. Efficacy and Safety of Intravitreal Aflibercept Treat-and-Extend Regimens in the ALTAIR Study: 96-Week Outcomes in the Polypoidal Choroidal Vasculopathy Subgroup. Adv Ther. 2022 Jun;39(6):2984-2998. doi: 10.1007/s12325-022-02162-w. Epub 2022 May 3. PMID 35503499
- [Derived] Ohji M, Okada AA, Sasaki K, Moon SC, Machewitz T, Takahashi K; ALTAIR Investigators. Relationship between retinal fluid and visual acuity in patients with exudative age-related macular degeneration treated with intravitreal aflibercept using a treat-and-extend regimen: subgroup and post-hoc analyses from the ALTAIR study. Graefes Arch Clin Exp Ophthalmol. 2021 Dec;259(12):3637-3647. doi: 10.1007/s00417-021-05293-y. Epub 2021 Jul 20. PMID 34283294
- [Derived] Ohji M, Takahashi K, Okada AA, Kobayashi M, Matsuda Y, Terano Y; ALTAIR Investigators. Efficacy and Safety of Intravitreal Aflibercept Treat-and-Extend Regimens in Exudative Age-Related Macular Degeneration: 52- and 96-Week Findings from ALTAIR : A Randomized Controlled Trial. Adv Ther. 2020 Mar;37(3):1173-1187. doi: 10.1007/s12325-020-01236-x. Epub 2020 Feb 3. PMID 32016788

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study was conducted in Japan between 19 December 2014 (first participant first visit) and 08 November 2017 (last participant last visit).
Pre-assignment Details: 288 participants were enrolled and 255 entered run-in phase. 8 were randomization failures. 247 participants were randomized (2 Weeks [2W] adjustment group: 124; 4 Weeks [4W] adjustment group: 123) at Week 16. All 247 participant:s were treated and 227 participants (111 in the 2W adjustment, 116 in the 4W adjustment) completed Week 52 treatment.
Groups:
- 2 Weeks Adjustment: Participants received Aflibercept Intravitreal (IVT) injection at Week 0, Week 4, Week 8 and Week 16 followed by the variable treatment intervals with the criteria of Treat and Extend regimen. In the case the study eye of a participant met the criteria, the length of treatment interval was to be extended or shortened by 2 weeks from the last interval, respectively. Minimum/Maximum treatment interval is 8 weeks and 16 weeks during Week 16 to 96.
- Randomization Failure: Participants entered run-in phase but discontinued the study before randomization after receiving at least one injection.
Period: Overall Study
Arm/Group | 2 Weeks Adjustment | 4 Weeks Adjustment | Randomization Failure
Started | 124 | 123 | 8
Treated | 124 | 123 | 7
Randomized | 124 | 123 | 0
BCVA Post-randomization Assessment | 123 | 123 | 0
Completed (Completed Treatment (Week 96)) | 108 | 104 | 0
Not Completed | 16 | 19 | 8
Not completed — Death | 2 | 1 | 0
Not completed — Progressive disease | 4 | 4 | 0
Not completed — Logistical difficulties | 1 | 3 | 0
Not completed — Protocol Violation | 0 | 3 | 0
Not completed — Physician Decision | 2 | 1 | 0
Not completed — Adverse Event | 4 | 2 | 0
Not completed — Withdrawal by Subject | 3 | 4 | 0
Not completed — Randomized failure | 0 | 0 | 8
Not completed — Required procedure failed | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: Safety analysis set (SAF): included all subjects who received any study drug
Groups:
- Total: Total of all reporting groups
Arm/Group | 2 Weeks Adjustment | 4 Weeks Adjustment | Randomization Failure | Total
Number analyzed (Participants) | 124 | 123 | 7 | 254
Age, Continuous [Mean (Standard Deviation); unit: years] | 73.0 (7.9) | 75.0 (8.1) | 80.3 (7.8) | 74.2 (8.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 36 | 32 | 1 | 69
  Male | 88 | 91 | 6 | 185
Best-corrected visual acuity (BCVA) [Mean (Standard Deviation); unit: letters] — Visual functions of the study eye at Screening screening visit were assessed, according to the Early Treatment Diabetic Retinopathy Study (ETDRS) protocol as described in detail in the operation manual.
  letters | 54.6 (13.1) | 55.3 (12.0) | 54.9 (17.9) | 55.0 (12.7)
Central Retinal Thickness [Mean (Standard Deviation); unit: μm] — Population: Participants in SAF with data available for central retinal thickness
  μm
    number analyzed (Participants) | 123 | 121 | 7 | 251
    (all) | 386.5 (158.6) | 370.3 (120.0) | 371.6 (88.5) | 378.3 (139.4)
Choroidal neovascularization [Count of Participants; unit: Participants]
  No CNV | 0 | 1 | 0 | 1
  Classic CNV | 35 | 42 | 1 | 78
  Classic & Occult | 15 | 17 | 2 | 34
  Occult | 72 | 62 | 4 | 138
  Unknown | 2 | 1 | 0 | 3
Typical age-related macular degeneration [Count of Participants; unit: Participants]
  Missing | 2 | 0 | 0 | 2
  No | 46 | 48 | 2 | 96
  Yes | 76 | 75 | 5 | 156
Polypoidal Choroidal Vasculopathy [Count of Participants; unit: Participants]
  Missing | 2 | 0 | 0 | 2
  No | 76 | 79 | 5 | 160
  Yes | 46 | 44 | 2 | 92
Retinal Angiomatous Proliferation [Count of Participants; unit: Participants]
  Missing | 2 | 0 | 0 | 2
  No | 118 | 114 | 6 | 238
  Yes | 4 | 9 | 1 | 14

OUTCOME MEASURES:

1. Primary Outcome: Mean Change From Baseline in BCVA at Week 52
Description: Visual functions of the study eye (at every visit) and the fellow eye were assessed, according to the ETDRS protocol as described in detail in the operation manual. A higher score represents better functioning.
Time Frame: Baseline and Week 52
Population: The outcome measure is analyzed based on full analysis set (FAS) including all randomized participants who received any study drug after randomization and had a baseline and at least one BCVA assessment after Week 16 (i.e. post randomization). The FAS was analyzed as randomized.
Measure: Mean (Standard Deviation); unit: letters
Arm/Group | 2 Weeks Adjustment | 4 Weeks Adjustment
Number analyzed (Participants) | 123 | 123
letters | 9.0 (14.6) | 8.4 (13.4)
Statistical Analysis 1: Comparison: 2 Weeks Adjustment vs 4 Weeks Adjustment; Test type: Superiority or Other; Least Square (LS) mean difference = -0.4, 95% CI 2-sided [-3.8 to 3.0]

2. Secondary Outcome: Percentage of Participants Who Maintained Vision at Week 52
Description: A participant was classified as maintaining vision if the participant had lost fewer than 15 letters in the ETDRS letter score compared to baseline.
Time Frame: Week 52
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | 2 Weeks Adjustment | 4 Weeks Adjustment
Number analyzed (Participants) | 123 | 123
percentage of participants | 96.7 [93.6 to 99.9] | 95.9 [92.4 to 99.4]
Statistical Analysis 1: Comparison: 2 Weeks Adjustment vs 4 Weeks Adjustment; Test type: Superiority or Other; Mantel-Haenszel (MH) adjusted difference = -0.9, 95% CI 2-sided [-5.7 to 4.0]

3. Secondary Outcome: Percentage of Participants Who Gained at Least 15 Letters of Vision Compared to Baseline at Week 52
Time Frame: Baseline and Week 52
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | 2 Weeks Adjustment | 4 Weeks Adjustment
Number analyzed (Participants) | 123 | 123
percentage of participants | 32.5 [24.2 to 40.8] | 30.9 [22.7 to 39.1]
Statistical Analysis 1: Comparison: 2 Weeks Adjustment vs 4 Weeks Adjustment; Test type: Superiority or Other; MH adjusted difference = -1.4, 95% CI 2-sided [-12.7 to 9.8]

4. Secondary Outcome: Mean Change in Central Retinal Thickness (CRT) From Baseline at Week 52
Time Frame: Baseline and week 52
Population: The outcome measure is analyzed based on full analysis set (FAS) with number of subjects evaluable for this specific end point.
Measure: Mean (95% Confidence Interval); unit: μm
Arm/Group | 2 Weeks Adjustment | 4 Weeks Adjustment
Number analyzed (Participants) | 123 | 123
μm | -134.4 [-162.2 to -106.6] | -126.1 [-147.1 to -105.1]
Statistical Analysis 1: Comparison: 2 Weeks Adjustment vs 4 Weeks Adjustment; Test type: Superiority or Other; LS mean difference = -5.8, 95% CI 2-sided [-24.3 to 12.7]

5. Secondary Outcome: Percentage of Participants Without Fluid on Optical Coherence Tomography (OCT) at Week 52
Description: A participant was classified as without fluid if "Evidence of new or persistent fluid" on OCT was "No".
Time Frame: Week 52
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | 2 Weeks Adjustment | 4 Weeks Adjustment
Number analyzed (Participants) | 123 | 123
Percentage of participants | 68.3 [60.1 to 76.5] | 69.1 [60.9 to 77.3]
Statistical Analysis 1: Comparison: 2 Weeks Adjustment vs 4 Weeks Adjustment; Test type: Superiority or Other; MH adjusted difference = 1.0, 95% CI 2-sided [-10.6 to 12.7]

ADVERSE EVENTS:
Time Frame: Up to 96 weeks
Arm/Group | 2 Weeks Adjustment | 4 Weeks Adjustment | Randomization Failure
Serious Adverse Events (participants affected / at risk) | 19/124 | 20/123 | 3/7
Other Adverse Events (participants affected / at risk) | 49/124 | 61/123 | 4/7
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | 2 Weeks Adjustment (N=124) | 4 Weeks Adjustment (N=123) | Randomization Failure (N=7)
Acute myocardial infarction (Cardiac disorders) | 0 | 1 | 0
Angina pectoris (Cardiac disorders) | 0 | 1 | 0
Angina unstable (Cardiac disorders) | 1 | 0 | 0
Coronary artery stenosis (Cardiac disorders) | 0 | 1 | 0
Tachycardia (Cardiac disorders) | 0 | 1 | 0
Sinus node dysfunction (Cardiac disorders) | 0 | 1 | 0
Cataract (Eye disorders) | 4 | 5 | 0
Age-related macular degeneration (Eye disorders) | 1 | 0 | 0
Gastric polyps (Gastrointestinal disorders) | 1 | 0 | 0
Ileus (Gastrointestinal disorders) | 0 | 1 | 0
Gastric mucosal lesion (Gastrointestinal disorders) | 0 | 1 | 0
Vascular stent stenosis (General disorders) | 0 | 1 | 0
Cholangitis (Hepatobiliary disorders) | 1 | 0 | 0
Cholecystitis (Hepatobiliary disorders) | 1 | 0 | 0
Cholecystitis acute (Hepatobiliary disorders) | 0 | 0 | 1
Cholelithiasis (Hepatobiliary disorders) | 2 | 1 | 0
Hepatic failure (Hepatobiliary disorders) | 0 | 1 | 0
Cellulitis (Infections and infestations) | 0 | 1 | 0
Diverticulitis (Infections and infestations) | 0 | 1 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 2
Vestibular neuronitis (Infections and infestations) | 1 | 0 | 0
Facial bones fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Femur fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Snake bite (Injury, poisoning and procedural complications) | 0 | 1 | 0
Spinal fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Spinal column stenosis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Bile duct cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 0
Laryngeal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Squamous cell carcinoma of lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Colon adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Gingival cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Dizziness (Nervous system disorders) | 0 | 1 | 0
Haemorrhage intracranial (Nervous system disorders) | 1 | 0 | 0
Hepatic encephalopathy (Nervous system disorders) | 0 | 1 | 0
Spinal epidural haematoma (Nervous system disorders) | 0 | 1 | 0
Nephrolithiasis (Renal and urinary disorders) | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | 2 Weeks Adjustment (N=124) | 4 Weeks Adjustment (N=123) | Randomization Failure (N=7)
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 1
Vertigo (Ear and labyrinth disorders) | 0 | 3 | 0
Cataract (Eye disorders) | 5 | 10 | 0
Conjunctival haemorrhage (Eye disorders) | 4 | 8 | 0
Dry eye (Eye disorders) | 3 | 6 | 0
Retinal pigment epithelial tear (Eye disorders) | 4 | 0 | 0
Age-related macular degeneration (Eye disorders) | 2 | 4 | 0
Constipation (Gastrointestinal disorders) | 4 | 7 | 0
Gastric ulcer (Gastrointestinal disorders) | 3 | 0 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 | 3 | 0
Nausea (Gastrointestinal disorders) | 3 | 1 | 0
Toothache (Gastrointestinal disorders) | 1 | 1 | 1
Large intestine polyp (Gastrointestinal disorders) | 0 | 4 | 0
Oedema peripheral (General disorders) | 1 | 1 | 1
Cholecystitis acute (Hepatobiliary disorders) | 0 | 0 | 1
Conjunctivitis (Infections and infestations) | 3 | 5 | 0
Influenza (Infections and infestations) | 2 | 4 | 0
Nasopharyngitis (Infections and infestations) | 26 | 20 | 0
Contusion (Injury, poisoning and procedural complications) | 1 | 4 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 3 | 0
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 3 | 0
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 | 3 | 0
Insomnia (Psychiatric disorders) | 3 | 1 | 0
Hypertension (Vascular disorders) | 1 | 4 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No